CLINICAL TRIAL: NCT00605878
Title: Studies of Skin Microflora in Healthy Individuals and Atopic Dermatitis Patients
Brief Title: Studies of Skin Microbes in Healthy People and in People With Skin Conditions
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080059; 08-HG-0059
Record Dates: First submitted 2008-01-23; First posted 2008-01-31 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-19

CONDITIONS: Eczema; Atopic Dermatitis
Keywords: Skin; Natural History; Microbiome; Bacteria; Atopic Dermatitis (Eczema); Atopic Dermatitis; Eczema; Health Volunteer; HG
MeSH Terms: conditions — Eczema; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Grouo 3: Healthy (pediatric) controls
- Group 1: Healthy (adult) volunteers
- Group 2: AD patients
- Group 4: Patients diagnosed with the primary immunodeficiency hyperIgE syndrome (HIES)
- Group 5: Patients diagnosed with the primary immunodeficiency Wiskott-Aldrich Syndrome (WAS)
- Group 6: Patients diagnosed with the combined immunodeficiency associated with DOCK8 mutation (DOCK8)

SUMMARY:
This study will examine microbes (e.g., bacteria, fungi, viruses) that live on human skin and how microbes contribute to health and disease. It will analyze healthy human skin and how the these microorganisms might change in patients with atopic dermatitis (AD), a skin condition also known as eczema.

Healthy volunteers, as well as patients with moderate to severe eczema (AD), between 2 and 40 years of age may be eligible for this study.

We also wish to enroll children and adults aged 2-40 who have been diagnosed with inherited immune disorders known as HIES (hyperimmunoglobulin-E syndrome), WAS (Wiskott-Aldrich syndrome), or DOCK8 immunodeficiency because they frequently have skin problems similar to AD.

Eligible participants undergo the following tests and procedures:

* Medical family and medication history
* Skin examination
* Blood tests (research blood as well as serum IgE, and complete blood count)
* Skin samples to analyze microbes. Samples are obtained by the following methods: swabbing the skin with a cotton swab; scraping (scratching) the skin gently with a blade to remove only the outermost skin layers; and, only in adults, biopsy (surgical removal) of a small skin sample less than 1/4-inch (5 mm) in diameter.
* Nose swabs to analyze microbes.
* Patients with eczema may have photographs of their skin taken to help monitor the skin rashes.

Participants may be contacted periodically for follow-up studies. Patients with atopic dermatitis may have additional skin samples collected to examine changes in the skin bacteria over time and during all of the stages of eczema. In addition, patients who have a flare of their eczema are asked to undergo a skin sample collection as soon as possible.

DETAILED DESCRIPTION:
* Skin microbiota (bacteria, fungi, viruses, phage, archae) play a significant role in common dermatological conditions, such as atopic dermatitis/AD (eczema).
* Since culture-dependent methods are often biased assessments of microbial diversity, genomic methods can expand our understanding of the human microbiome and skin diseases.
* Chronic dermatitis is typical among rare primary immunodeficiencies: Wiskott-Aldrich syndrome; hyper-IgE syndrome; and combined immunodeficiency associated with DOCK8 mutation syndrome. The skin disease in these monogenic disorders resembles AD, is associated with microbial infections, and may provide additional insight into microbial-host disease interactions.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for all groups

Must have a primary care professional who will continue standard of care/evaluation in tandem with the protocol to whom information and recommendations can be communicated.

Inclusion Criteria for Group 1: Healthy Volunteers

Adult males or females aged 18-50 at time of enrollment.

Inclusion Criteria for Group 2: AD patients

A. Confirmed diagnosis of AD (UK Working Party s Diagnostic Criteria)24

B. Moderate to severe AD SCORAD greater than or equal to 25(25)

C. Greater than or equal to 1 affected antecubital (or popliteal) fossae at time of enrollment to serve as a target site.

Inclusion Criteria for Group 3: Healthy (pediatric) Controls

A. Males or females 2-18 years of age.

Inclusion Criteria for Groups 4, 5, & 6: AD/HIES/WAS/DOCK8 patients

A. Must have mutation-proven diagnosis, with or without eczematous dermatitis.

EXCLUSION CRITERIA:

Exclusion Criteria for all groups:

1. Any subjects receiving or planning to receive an IND agent, ultraviolet light therapy, monoclonal antibodies, or systemic immunosuppressants < 7 days or 5 half-lives (whichever is the longer time period) of initiating this protocol.
2. Any subjects who have cancer, and are currently or have previously received treatment with chemotherapy or radiation for treatment of malignancies within the previous 6 months.
3. Any subject with a history of bone marrow transplant or gene therapy.

Exclusion Criteria specific for Group 2: AD patients

A. Unable to remain off systemic (oral) antibiotics or systemic (oral) steroids for at least 7 days prior to body site sampling. Unable to temporarily discontinue use of topical steroids or calcineurin inhibitors for greater than or equal to 7 days to small areas of skin intended for sampling. (Topical therapies/emollients for AD may be continued to non-adjacent, nontarget sites.)

B. Underlying immunodeficiency, either as primary disease or secondary to treatment.

Exclusion Criteria specific for Groups 4, 5, & 6: HIES/WAS/DOCK8 patients:

A. Unable to remain off topical steroids and emollients for preferably 7 days but at least 24 hours prior to body site sampling.

Exclusion Criteria specific for Groups 1 & 3: Healthy Volunteers and Healthy (pediatric) Controls:

A. Any subjects with unstable or uncontrolled or chronic medical conditions requiring treatment or hospitalization. Individual determinations will be made at the discretion of the medical investigator.

B. Underlying immunodeficiency, either as primary disease or secondary to treatment.

C. Other documented chronic dermatologic disease, such as AD or psoriasis that may interfere with evaluation of the cutaneous microbiome. Common transient conditions, such as acne, are permissible.

D. Subjects who provide direct healthcare or reside in healthcare facilities or in non-hospital settings such as assisted living facilities, homeless shelters, jails and prisons as well as subjects with frequent exposure to laboratory animals.

E. Subjects with asthma.

5. Any female with symptoms and/or serum hormone levels consistent with perimenopause

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy (adult) volunteers AD patients Healthy (pediatric) controls Patients diagnosed with the primary immunodeficiency hyperIgE syndrome (HIES) Patients diagnosed with the primary immunodeficiency Wiskott-Aldrich Syndrome (WAS) Patients diagnosed with the combined immunodeficiency associated with DOCK8 mutation (DOCK8)
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2008-01-22 (Actual)

PRIMARY OUTCOMES:
Primary Immunodeficiency | Ongoing
  Analyze the microbiome of patients with primary immunodeficiency disorders that are known to have AD-like skin disease.
Healthy volunteers | Ongoing
  Characterize the microbiome of healthy individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Segre, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oh J, Freeman AF; NISC Comparative Sequencing Program; Park M, Sokolic R, Candotti F, Holland SM, Segre JA, Kong HH. The altered landscape of the human skin microbiome in patients with primary immunodeficiencies. Genome Res. 2013 Dec;23(12):2103-14. doi: 10.1101/gr.159467.113. Epub 2013 Oct 29. PMID 24170601
- [Background] Oh J, Byrd AL, Deming C, Conlan S; NISC Comparative Sequencing Program; Kong HH, Segre JA. Biogeography and individuality shape function in the human skin metagenome. Nature. 2014 Oct 2;514(7520):59-64. doi: 10.1038/nature13786. PMID 25279917
- [Background] Gao Z, Tseng CH, Pei Z, Blaser MJ. Molecular analysis of human forearm superficial skin bacterial biota. Proc Natl Acad Sci U S A. 2007 Feb 20;104(8):2927-32. doi: 10.1073/pnas.0607077104. Epub 2007 Feb 9. PMID 17293459
- [Derived] Ahmed N, Joglekar P, Deming C; NISC Comparative Sequencing Program; Lemon KP, Kong HH, Segre JA, Conlan S. Genomic characterization of the C. tuberculostearicum species complex, a prominent member of the human skin microbiome. mSystems. 2023 Dec 21;8(6):e0063223. doi: 10.1128/msystems.00632-23. Epub 2023 Nov 10. PMID 38126779
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2008-HG-0059.html